CLINICAL TRIAL: NCT04964206
Title: Impact of Maternal Neuraxial Labor Analgesia on Offspring Neurodevelopment. A Multicenter, Prospective, Longitudinal Cohort Study
Brief Title: Neuraxial Labor Analgesia and Offspring Neurodevelopment
Status: Recruiting | Type: Observational
Sponsor: Dong-Xin Wang (Other)
Collaborators: Shenzhen Maternity and Child Healthcare Hospital (Unknown)
Responsible Party: Sponsor-Investigator, Dong-Xin Wang, Professor and Chairman, Department of Anesthesiology and Critical Care Medicine, Peking University First Hospital
Organization: Peking University First Hospital (Other)
Other Study IDs: 2021-026
Record Dates: First submitted 2021-07-06; First posted 2021-07-16 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Offspring, Adult; Labor Pain; Maternal Anesthesia and Analgesia Affecting Fetus or Newborn; Neurodevelopmental Delay; Postpartum Depression
Keywords: Neuraxial labour analgesia; Neurodevelopmental delay
MeSH Terms: conditions — Labor Pain; Depression, Postpartum

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Neuraxial analgesia exposure: For mothers who accept neuraxial labor analgesia, epidural analgesia or combined spinal-epidural analgesia will be provided according to routine practice of each study center.
  Interventions: Procedure: Neuraxial labor analgesia
- No neuraxial analgesia exposure: For patients who do not accept neuraxial labor analgesia, analgesics will be prescribed by obstetricians according to routine practice.
  Interventions: Procedure: No neuraxial labor analgesia

INTERVENTIONS:
Procedure: Neuraxial labor analgesia — Epidural or combined spinal-epidural labor analgesia will be performed according to the routine practice of each study center.
  Groups: Neuraxial analgesia exposure
Procedure: No neuraxial labor analgesia — Neuraxial analgesia will not be performed. Analgesics will be prescribed by the obstetricians according to routine practice.
  Groups: No neuraxial analgesia exposure

SUMMARY:
How perinatal factors affect the long-term development of children has always been an issue of much concern. This study is designed to explore the potential impact of maternal neuraxial labor analgesia exposure on offspring neurodevelopment.

DETAILED DESCRIPTION:
Neuraxial labor analgesia, including epidural analgesia and combined spinal-epidural analgesia, is a well-established technique to alleviate labor pain. It can help to reduce the maternal stress response during labor and might be associated with a lower risk of maternal postpartum depression; which may be beneficial to the long-term neurodevelopment in offspring.

On the other hand, neuraxial labor analgesia is associated with increased risks of intrapartum maternal fever and instrumental delivery, which may produce potentially harmful effects. In addition, it has been reported that the anesthetic exposure during neuraxial analgesia may lead to fetal-neonatal depression and even neurotoxic effects of less mature neonatal brain. Taking all these into account, the potential long-term effects of neuraxial analgesia on offspring neurodevelopment is still controversial and deserves further study.

The objective of study is to investigate if there is any association between maternal neuraxial analgesia exposure during labor and risk of offspring neurodevelopment delay at age 24 months.

ELIGIBILITY:
Inclusion Criteria:

1. Primiparae between 18 and 35 years of age with term single cephalic pregnancy;
2. Undergo regular prenatal examination in the study centers;
3. Preparing to deliver vaginally.

Exclusion Criteria:

1. History of psychiatric diseases (indicate those that are diagnosed before or during pregnancy by psychiatrists);
2. History of diseases involving the hypothalamic-pituitary-adrenal axis;
3. Presence of contraindications to epidural analgesia, which includes: (1) History of infectious disease of the central nervous system (poliomyelitis, cerebrospinal meningitis, encephalitis, etc.); (2) History of spinal or intra-spinal disease (trauma or surgery of spinal column, intra-spinal canal mass, etc.); (3) Systemic infection (sepsis); (4) Skin or soft tissue infection at the site of epidural puncture; (5) Coagulopathy.
4. Presence of contraindications to vaginal delivery;
5. Other reasons that are considered unsuitable for study participation.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Primiparae between 18 and 35 years of age with term single cephalic pregnancy who undergo regular prenatal examination in the study centers and are preparing to deliver vaginally.
Sampling Method: Non-Probability Sample
Enrollment: 5580 (Estimated)
Dates: Start 2022-10-14 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of developmental delay in offspring at 24 months of age | At 24 months of age
  The Ages & Stages Questionnaires® in Chinese, 3rd edition (ASQ®-3 Chinese) will be used to detect developmental delays among children from 1 month to 60 months of age. The ASQ®-3 Chinese contains 30 items representing five developmental domains: communication, gross motor, fine motor, problem solving, and personal-social behavior. For each domain, a score that is more than 2 standard deviations below the mean indicates suspected developmental delay. A score below the threshold in any of the 5 domains indicates suspected developmental delay.

SECONDARY OUTCOMES:
Incidence of developmental delay in offspring at 6 and 12 months of age | At 6 and 12 months of age
  The Ages & Stages Questionnaires® in Chinese, 3rd edition (ASQ®-3 Chinese) will be used to detect developmental delays among children from 1 month to 60 months of age. The ASQ®-3 Chinese contains 30 items representing five developmental domains: communication, gross motor, fine motor, problem solving, and personal-social behavior. For each domain, a score that is more than 2 standard deviations below the mean indicates suspected developmental delay. A score below the threshold in any of the 5 domains indicates suspected developmental delay.
Maternal intrapartum fever | Up to the end of childbirth (stage 3)
  Defined as the highest maternal temperature ≥38.0℃ during any stage of labor.
Neonatal Apgar score <8 at 1 and 5 minutes after delivery | At 1 and 5 minutes after delivery
  Neonatal Apgar score is assessed and recorded by gynecologists or midwives at 1 and 5 minutes after delivery.
Histologic chorioamnionitis | Up to hospital discharge
  According to pathological examination of placenta
Neonatal infection | Within 3 days after birth
  Neonatal infection is defined by the occurrence of 1 or more of the following: neonatal sepsis, neonatal uncharacterized infection, neonatal pneumonia, or neonatal necrotizing enterocolitis diagnosed according to the Chinese Classification of Disease and Codes (Version 2.0, International Statistical Classification of Diseases and Related Health Problems, Tenth Revision [ICD-10]) established by the Chinese government.
Depression score of mothers | At 42 days, 6 months, 12 months, and 24 months after childbirth
  Maternal depression is assessed with the Edinburgh Postnatal Depression Scale. A score of 10 or higher is defined the presence of depressive symptoms.

OTHER OUTCOMES:
Use of oxytocin | Up to the end of childbirth (stage 3)
  Use of oxytocin during the intrapartum period.
Maternal use of antibiotics | Up to hospital discharge
  Maternal use of antibiotics
Neonatal admission to the neonatal intensive care unit | Up to hospital discharge
  Neonatal admission to the neonatal intensive care unit
Neonatal use of antibiotics | Up to hospital discharge
  Neonatal use of antibiotics
Persistent pain | At 42 days postpartum
  Persistent or recurrent pain that lasted for more than 1 months after childbirth.
Covid-19 infection | During pregnancy
  Covid-19 related information was collect before delivery, including whether participants were infected, during pregnancy, what covid-19 related symptoms they had, whether participants received covid-19 vaccine. Performed in part of enrolled patients.

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Xin Wang, MD,PHD, Principal Investigator — Peking University First Hospital
Locations (2):
- China (2):
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Shenzhen Maternity and Child Healthcare Hospital, Shenzhen, Guangdong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Liu ZH, He ST, Deng CM, Ding T, Xu MJ, Wang L, Li XY, Wang DX. Neuraxial labour analgesia is associated with a reduced risk of maternal depression at 2 years after childbirth: A multicentre, prospective, longitudinal study. Eur J Anaesthesiol. 2019 Oct;36(10):745-754. doi: 10.1097/EJA.0000000000001058. PMID 31356375
- [Background] Wong CA. Advances in labor analgesia. Int J Womens Health. 2010 Aug 9;1:139-54. doi: 10.2147/ijwh.s4553. PMID 21072284
- [Background] Morton S, Kua J, Mullington CJ. Epidural analgesia, intrapartum hyperthermia, and neonatal brain injury: a systematic review and meta-analysis. Br J Anaesth. 2021 Feb;126(2):500-515. doi: 10.1016/j.bja.2020.09.046. Epub 2020 Nov 18. PMID 33218673
- [Background] Flick RP, Lee K, Hofer RE, Beinborn CW, Hambel EM, Klein MK, Gunn PW, Wilder RT, Katusic SK, Schroeder DR, Warner DO, Sprung J. Neuraxial labor analgesia for vaginal delivery and its effects on childhood learning disabilities. Anesth Analg. 2011 Jun;112(6):1424-31. doi: 10.1213/ANE.0b013e3181f2ecdd. Epub 2010 Aug 24. PMID 20736436
- [Background] Wall-Wieler E, Bateman BT, Hanlon-Dearman A, Roos LL, Butwick AJ. Association of Epidural Labor Analgesia With Offspring Risk of Autism Spectrum Disorders. JAMA Pediatr. 2021 Jul 1;175(7):698-705. doi: 10.1001/jamapediatrics.2021.0376. PMID 33871547
- [Background] Wei M, Bian X, Squires J, Yao G, Wang X, Xie H, Song W, Lu J, Zhu C, Yue H, Zhu G, Wang Q, Xu R, Wan C, Sun S, Chen J. [Studies of the norm and psychometrical properties of the ages and stages questionnaires, third edition, with a Chinese national sample]. Zhonghua Er Ke Za Zhi. 2015 Dec;53(12):913-8. Chinese. PMID 26887546